CLINICAL TRIAL: NCT05897359
Title: The Use of Nursing-students-led bCBTMI for Internet Addiction Among Adolescents: a Feasibility Cluster Randomised Controlled Trial
Brief Title: The Use of Nursing-students-led bCBTMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Katherine Lam, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bCBTMI-Adolescents
Record Dates: First submitted 2023-05-11; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Internet Addiction
Keywords: Adolescents; Nursing-students-led; Cognitive Behavioural therapy; Motivational Interviewing
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bCBTMI (Experimental): bCBTMI care for IA.
  Interventions: Behavioral: bCBTMI
- Control (Placebo Comparator): Routine care for IA.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: bCBTMI — This experimental group involves 4 weekly 30-45 minute sessions using the brief CBT and the brief MI models by trained nursing students.
  Arms: bCBTMI
Behavioral: Control — The control group will receive health talks about internet addiction consequences and impacts on young people by nursing students who are not involved in the intervention group to mimic the time and attention spent on the intervention group. These health talks are considered routine care for IA health promotion.
  Arms: Control

SUMMARY:
The use of the internet is very popular in adolescence. Notwithstanding the benefits from the internet, many users are addicted to the internet and develop problematic behaviours which are regarded as "Internet addiction" (IA). Trained nursing students, who are the future nurses and well-equipped with basic health knowledge, as the interventionists to deliver a bCBTMI intervention to the eligible subjects. The result of this study is expected to provide evidence of the feasibility and effectiveness of training nursing students to conduct bCBTMI in Hong Kong Chinese adolescents with IA for a definitive RCT.

DETAILED DESCRIPTION:
A two-arm, parallel-group, feasibility cluster randomized controlled trial will be conducted. 60 adolescents with IA will be recruited from secondary schools in Hong Kong. Participants in the intervention group will receive 4 weekly 30-45 minute sessions using the brief CBT and the brief MI models by nursing students. Control group participants will receive routine care for IA.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13 to 17
* Studying Forms 2 to 4
* Classified as IA by the Chinese version of Young's 10-item Internet Addiction Test (IAT)
* Can communicate in Cantonese and read Chinese.

Exclusion Criteria:

* With physical or cognitive impairment and learning problems as identified from the medical records

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Screening rate | at day 1
  Calculated as the number of students screened at participated secondary schools divided by number of students at participated schools during the recruitment period.
Eligibility rate | at day 1
  Calculated by dividing the number of secondary school students who are eligible by the number who are screened.
Consent rate | at the 6-month follow-up
  Calculated by dividing the number of secondary school students who consent to join the study by the number who are eligible.
Randomization rate | at day 1
  Calculated by dividing the number of secondary school students who are randomized into intervention and control groups by those who provide consent.
Attendance rate | Immediately after the bCBTMI intervention
  Calculated by dividing the number of secondary school students who complete the intervention by those who are randomized.
Retention rate | at the 6-month follow-up
  Calculated by dividing the number of secondary school students who remain in the study by those who are randomized. Retention rates for the intervention and control groups will be calculated at each follow-up.
Adherence to intervention protocol | at the 1-month follow-up
  Calculated by dividing the number of secondary school students who follow the intervention protocol by those who are randomized.
Complete rate | at the 6-month follow-up
  Calculated by dividing the number of secondary school students who returned questionnaires by the number of questionnaires distributed. This will be calculated by groups at baseline and each follow-up.
Missing data | at the 6-month follow-up
  Calculated as the percentage of missing values in the dataset. Unknown or blank values will be considered missing values.
Adverse events | at the 6-month follow-up
  Are defined as unfavorable and unintended events that are not present at baseline, or appear to have worsened during the study. The relation to the intervention will be assessed in accordance with the protocol for adverse events management (It can be provided upon request). The number and event severity will be recorded. Numbers and reasons for exclusions will be noted.

SECONDARY OUTCOMES:
Self-reported abstinence at the 1-week follow-up | at the 1-week follow-up
  Measured by the number of IA symptoms via a self-reported questionnaire.
Self-reported abstinence at the 1-month follow-up | at the 1-month follow-up
  Measured by the number of IA symptoms via a self-reported questionnaire.
Self-reported abstinence at the 3-month follow-up | at the 3-month follow-up
  Measured by the number of IA symptoms via a self-reported questionnaire.
Self-reported abstinence at the 6-month follow-up | at the 6-month follow-up
  Measured by the number of IA symptoms via a self-reported questionnaire.
The Chinese version of Center for Epidemiologic Studies Depression Scale for Children (CES-DC) | at the 1-week follow-up
  CES-DC will be used to record the number of depression symptoms in secondary schools students with IA at each follow-up. It includes 20 items asking on a 4-point Likert scale in relation to the incidence of the stated symptoms during the previous week, and are scored from 0 to 3 (0 = not at all, 3 = a lot). Total scores range from 0 to 60, with higher scores indicating greater number of depressive symptoms. This questionnaire has been empirically tested and validated in Hong Kong children and are currently using in Youth Quitline.
The Chinese version of Center for Epidemiologic Studies Depression Scale for Children (CES-DC) | at the 1-month follow-up
  CES-DC will be used to record the number of depression symptoms in secondary schools students with IA at each follow-up. It includes 20 items asking on a 4-point Likert scale in relation to the incidence of the stated symptoms during the previous week, and are scored from 0 to 3 (0 = not at all, 3 = a lot). Total scores range from 0 to 60, with higher scores indicating greater number of depressive symptoms. This questionnaire has been empirically tested and validated in Hong Kong children and are currently using in Youth Quitline.
The Chinese version of Center for Epidemiologic Studies Depression Scale for Children (CES-DC) | at the 3-month follow-up
  CES-DC will be used to record the number of depression symptoms in secondary schools students with IA at each follow-up. It includes 20 items asking on a 4-point Likert scale in relation to the incidence of the stated symptoms during the previous week, and are scored from 0 to 3 (0 = not at all, 3 = a lot). Total scores range from 0 to 60, with higher scores indicating greater number of depressive symptoms. This questionnaire has been empirically tested and validated in Hong Kong children and are currently using in Youth Quitline.
The Chinese version of Center for Epidemiologic Studies Depression Scale for Children (CES-DC) | at the 6-month follow-up
  CES-DC will be used to record the number of depression symptoms in secondary schools students with IA at each follow-up. It includes 20 items asking on a 4-point Likert scale in relation to the incidence of the stated symptoms during the previous week, and are scored from 0 to 3 (0 = not at all, 3 = a lot). Total scores range from 0 to 60, with higher scores indicating greater number of depressive symptoms. This questionnaire has been empirically tested and validated in Hong Kong children and are currently using in Youth Quitline.
Anxiety level | at the 1-week follow-up
  The anxiety level of secondary school students with IA will be measured by the short form of the Chinese Version of the State Anxiety Scale for Children (CSAS-C) at each follow-up. It has 10 itmes with scores from 1 to 3. Total scores range from 10 to 30, with higher scores indicating a higher level of anxiety. This questionnaire has been empirically tested and validated in Hong Kong children.
Anxiety level | at the 1-month follow-up
  The anxiety level of secondary school students with IA will be measured by the short form of the Chinese Version of the State Anxiety Scale for Children (CSAS-C) at each follow-up. It has 10 itmes with scores from 1 to 3. Total scores range from 10 to 30, with higher scores indicating a higher level of anxiety. This questionnaire has been empirically tested and validated in Hong Kong children.
Anxiety level | at the 3-month follow-up
  The anxiety level of secondary school students with IA will be measured by the short form of the Chinese Version of the State Anxiety Scale for Children (CSAS-C) at each follow-up. It has 10 itmes with scores from 1 to 3. Total scores range from 10 to 30, with higher scores indicating a higher level of anxiety. This questionnaire has been empirically tested and validated in Hong Kong children.
Anxiety level | at the 6-month follow-up
  The anxiety level of secondary school students with IA will be measured by the short form of the Chinese Version of the State Anxiety Scale for Children (CSAS-C) at each follow-up. It has 10 itmes with scores from 1 to 3. Total scores range from 10 to 30, with higher scores indicating a higher level of anxiety. This questionnaire has been empirically tested and validated in Hong Kong children.
Sleep quality of secondary schools students with IA will be assessed using the Pittsburgh Sleep Quality Index (PSQI) | at the 1-week follow-up
  It contains 19 items measuring 7 domains: subjective sleep quality, latency, duration, habitual efficiency, disturbances, use of medication, and daytime dysfunction on a 3-point scale (0: no difficulty to 3: severe difficulty) except for the items reporting bedtime and time awake. The sum of the seven component scores produces a global score with higher scores represent poorer subjective sleep quality. It has been validated in Hong Kong children and adolescents previously.
Sleep quality of secondary schools students with IA will be assessed using the Pittsburgh Sleep Quality Index (PSQI) | at the 1-month follow-up
  It contains 19 items measuring 7 domains: subjective sleep quality, latency, duration, habitual efficiency, disturbances, use of medication, and daytime dysfunction on a 3-point scale (0: no difficulty to 3: severe difficulty) except for the items reporting bedtime and time awake. The sum of the seven component scores produces a global score with higher scores represent poorer subjective sleep quality. It has been validated in Hong Kong children and adolescents previously.
Sleep quality of secondary schools students with IA will be assessed using the Pittsburgh Sleep Quality Index (PSQI) | at the 3-month follow-up
  It contains 19 items measuring 7 domains: subjective sleep quality, latency, duration, habitual efficiency, disturbances, use of medication, and daytime dysfunction on a 3-point scale (0: no difficulty to 3: severe difficulty) except for the items reporting bedtime and time awake. The sum of the seven component scores produces a global score with higher scores represent poorer subjective sleep quality. It has been validated in Hong Kong children and adolescents previously.
Sleep quality of secondary schools students with IA will be assessed using the Pittsburgh Sleep Quality Index (PSQI) | at the 6-month follow-up
  It contains 19 items measuring 7 domains: subjective sleep quality, latency, duration, habitual efficiency, disturbances, use of medication, and daytime dysfunction on a 3-point scale (0: no difficulty to 3: severe difficulty) except for the items reporting bedtime and time awake. The sum of the seven component scores produces a global score with higher scores represent poorer subjective sleep quality. It has been validated in Hong Kong children and adolescents previously.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Wai Katherine Lam, Principal Investigator — School of Nursing, Hong Kong Polytechnic University
Locations (1):
- Katherine Lam, Hong Kong, Hong Kong,China, Hong Kong